CLINICAL TRIAL: NCT06479967
Title: The Effects of Virtual Reality and Music on Pain, Anxiety, Itching, and Vital Signs During Skin Prick Testing: A Randomized Controlled Trial
Brief Title: The Effects of Virtual Reality and Music on Pain, Anxiety, Itching, and Vital Signs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, EDA UNAL, principal investigator, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EU13021985
Record Dates: First submitted 2024-05-13; First posted 2024-06-28 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Allergy; Anxiety; Pain; Itching; Vital Signs
Keywords: allergy; skin test; children; itching; musictherapy; Pain; Anxiety; Virtual Reality
MeSH Terms: conditions — Hypersensitivity; Anxiety Disorders; Pain; Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality (Experimental): The Virtual Reality glasses group watched a cartoon video of "Rafadan Tayfa Gizli Hazine" The VR glasses group watched a cartoon video of "Rafadan Tayfa Gizli Hazine" After the SPT, the VR glasses group took a 1-minute break from watching videos and the child's pain was assessed with WBFPS. During the 15-minute SPT assessment, the VR glasses group continued watching cartoon
  Interventions: Other: The VR glasses group
- Music (Experimental): The music group listened to classical piano "The Best of Chopin."
  After the music group took a 1-minute break from listening to music, and the child's pain was assessed with WBFPS. During the 15-minute SPT assessment, the music group continued to listen to the music. During the SPT evaluation, the music group took a 1-minute break from listening to music at 5, 10, and 15 minutes, and the child evaluated the level of itching from 1 to 10.
  Interventions: Other: the music group
- Control (No Intervention): Before, during, and after the skin prick test evaluation (15 minutes), no intervention was provided to the children assigned to the control group.

INTERVENTIONS:
Other: The VR glasses group — The Virtual Reality glasses group watched a cartoon video of "Rafadan Tayfa Gizli Hazine" The VR glasses group watched a cartoon video of "Rafadan Tayfa Gizli Hazine" After the SPT, the VR glasses group took a 1-minute break from watching videos and the child's pain was assessed with WBFPS. During the 15-minute SPT assessment, the VR glasses group continued watching cartoon
  Arms: Virtual Reality
Other: the music group — The music group listened to classical piano "The Best of Chopin." After the music group took a 1-minute break from listening to music, and the child's pain was assessed with WBFPS. During the 15-minute SPT assessment, the music group continued to listen to the music. During the SPT evaluation, the music group took a 1-minute break from listening to music at 5, 10, and 15 minutes, and the child evaluated the level of itching from 1 to 10.
  Arms: Music

SUMMARY:
Aim: This study aimed to examine the effects of virtual reality and music on pain, anxiety, itching, and vital signs of children during a skin prick test and evaluation.

Background:Virtual reality and music are utilised to reduce pain, anxiety, and itching in children throughout various treatment processes.

Methods: This randomised controlled trial was divided into three groups: Virtual reality (n=30), music (n=30), and control (n=30). Anxiety was assessed before and after the skin prick test using the "State-Trait Anxiety Inventory for Children"; pain was assessed during and after the skin prick test using the "Wong-Baker Faces Pain Rating Scale"; vital signs were measured before, during, and after the skin prick test, and the itch assessment "Visual Analogue Score" was assessed at 5, 10, and fifteen minutes after the skin prick test. The study followed the CONCORT guideline.

DETAILED DESCRIPTION:
The Effects of Virtual Reality and Music on Pain, Anxiety, Itching, and Vital Signs During Skin Prick Testing: A Randomized Controlled Trial ABSTRACT Aim: This study aimed to examine the effects of virtual reality and music on pain, anxiety, itching, and vital signs of children during a skin prick test and evaluation.

Background:Virtual reality and music are utilised to reduce pain, anxiety, and itching in children throughout various treatment processes.

Methods: This randomised controlled trial was divided into three groups: Virtual reality (n=30), music (n=30), and control (n=30). Anxiety was assessed before and after the skin prick test using the "State-Trait Anxiety Inventory for Children"; pain was assessed during and after the skin prick test using the "Wong-Baker Faces Pain Rating Scale"; vital signs were measured before, during, and after the skin prick test, and the itch assessment "Visual Analogue Score" was assessed at 5, 10, and fifteen minutes after the skin prick test. The study followed the CONCORT guideline.

Key words: allergy skin test, children, pain, anxiety, itching, virtual reality glasses, music.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 9-12 undergoing their initial skin test
* With no cognitive, visual, or auditory impairments
* No recent medical encounters involving pain or anxiety within the past 3 months
* Parents who volunteered for participation in this study.

Exclusion Criteria:

* Those who are not between the ages of 9 and 12 and have had a skin prick test before
* With cognitive, visual, or auditory impairments,
* Recent medical encounters involving pain or anxiety within the past 3 months,
* Parents who volunteered no for participation in this study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-11-12 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Anxiety level | 12 week
  State-Trait Anxiety Inventory for Children (minimum score of 20 and a maximum score of 60)
Pain Levels | 12 week
  Wong-Baker Faces Pain Rating Scale (a score of "0" to excruciating pain a value of "10")
Itching level | 12 week
  Visual Analogue Score ( rate the severity of the itch on a scale of one to ten) maximum 10axsimum 10
Heart Rate | 12 weeks
  Heart Rate ( pulse rate 70-110 ) ( /minute ) In the 9-12 age range, the lower pulse value is 70 and the upper value is 110.
Oxygen Saturation | 12 week
  Oxygen Saturation. ( between % 95-100)
Respiratory Rate | 12 weeks
  Respiratory Rate ( one minute ) (/minute). Between 16-22 / minute

CONTACTS AND LOCATIONS:
Overall Officials: Eda UNAL, PhD, Principal Investigator — Uludag universty; Aysel OZDEMIR, PhD, Study Director — Uludag University
Locations (1):
- Uludag Üniversty, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No.

REFERENCES:
- [Background] Baschong A, Spiess F, Cattin PC, Navarini A, Mueller SM. Itch reduction using immersive virtual reality-An experimental pilot study. Dermatol Ther. 2021 Jul;34(4):e15001. doi: 10.1111/dth.15001. Epub 2021 Jun 9. PMID 34036696
- [Background] da Silva Santa IN, Schveitzer MC, Dos Santos MLBM, Ghelman R, Filho VO. MUSIC INTERVENTIONS IN PEDIATRIC ONCOLOGY: Systematic review and meta-analysis. Complement Ther Med. 2021 Jun;59:102725. doi: 10.1016/j.ctim.2021.102725. Epub 2021 May 5. PMID 33964406
- [Background] Demirtas S, Houssais C, Tanniou J, Misery L, Brenaut E. Effectiveness of a music intervention on pruritus: an open randomized prospective study. J Eur Acad Dermatol Venereol. 2020 Jun;34(6):1280-1285. doi: 10.1111/jdv.16149. Epub 2020 Jan 14. PMID 31838780
- [Background] Goldberg A, Stauber T, Peleg O, Hanuka P, Eshayek L, Confino-Cohen R. Medical clowns ease anxiety and pain perceived by children undergoing allergy prick skin tests. Allergy. 2014 Oct;69(10):1372-9. doi: 10.1111/all.12463. Epub 2014 Aug 4. PMID 24943088